CLINICAL TRIAL: NCT07092384
Title: Effect of Remifentanil on Pruritus and Paresthesia Caused by Fospropofol Disodium Anesthesia
Brief Title: Effect of Remifentanil on Pruritus and Paresthesia of Fospropofol Disodium Anesthesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tongji Hospital (Other)
Responsible Party: Principal Investigator, aijun xu, Clinical Professor, Tongji Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ERPF
Record Dates: First submitted 2025-07-15; First posted 2025-07-29 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Remifentanil; Adverse Effects
MeSH Terms: interventions — Remifentanil; Sufentanil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Group R1 (Experimental): remifentanil 0.5μg/kg
  Interventions: Drug: Remifentanil
- Group R2 (Experimental): remifentanil 1.0μg/kg
  Interventions: Drug: Remifentanil
- Group R3 (Experimental): remifentanil 1.5μg/kg
  Interventions: Drug: Remifentanil
- Group R4 (Experimental): remifentanil 2.0μg/kg
  Interventions: Drug: Remifentanil
- Group S (Active Comparator): sufentanil 0.3μg/kg
  Interventions: Drug: Sufentanil

INTERVENTIONS:
Drug: Remifentanil — Observe the incidence of pruritus and paresthesia after different doses of remifentanil and fospropofol disodium
  Other Names: remi
  Arms: Group R1; Group R2; Group R3; Group R4
Drug: Sufentanil — Observe the incidence of pruritus and paresthesia after sufentanil and fospropofol disodium
  Other Names: sufen
  Arms: Group S

SUMMARY:
Explore the effect of remifentanil on pruritus and paresthesia induced by fospropofol disodium in adults

DETAILED DESCRIPTION:
Explore the effect of remifentanil on pruritus and paresthesia caused by fospropofol disodium in adults, to observe the manifestations and duration of pruritus and paresthesia

ELIGIBILITY:
Inclusion Criteria:

* Age 18-80 years old, plans to undergo elective non-cardiac surgery under general anesthesia.
* ASA I-II;
* The operation duration > 30 min;
* BMI 18-30kg /m2；
* Sign the informed consent form.

Exclusion Criteria:

* history of drug abuse or alcohol dependence;
* used sedative or analgesic drugs before operation;
* with severe liver and kidney function impairment;
* allergic to propofol and lipids;
* surgery that directly affect hemodynamics with surgical operations, such as macrovascular surgery;
* abnormal coagulation function, endocrine diseases or other effects on hemodynamic status;
* Participation in other clinical researchers in the past 3 months

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 265 (Actual)
Dates: Start 2025-07-30 (Actual); Primary Completion 2025-11-30 (Actual); Study Completion 2025-12-01 (Actual)

PRIMARY OUTCOMES:
Incidence of pruritus and paresthesia after administration of fospropofol disodium | 24 hours
  Observe the incidence of pruritus and paresthesia in patients within 3 minutes after administration

SECONDARY OUTCOMES:
Time of pruritus or paresthesia | 1 day
  time of pruritus and paresthesia occur after administration and 24h after surgery
dosage of drugs | 1 day
  Doses of drugs used during induction and maintenance of anesthesia
time records checklist | 1 day
  anesthesia time, induction time, surgical time, awakening time, and recovery time
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | 1 day
  Incidence of Treatment-Emergent Adverse Events
duration of pruritus or paresthesia | 24 hours
  pruritus and paresthesia occur after administration and 24h after surgery

CONTACTS AND LOCATIONS:
Overall Officials: aihua Du, Dr., Study Chair — Tongji Hospital
Locations (1):
- Tongji Hospital, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No